CLINICAL TRIAL: NCT05156411
Title: Strength Training With Eccentric Arm-cranking
Acronym: KREHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-26
Record Dates: First submitted 2021-11-08; First posted 2021-12-14 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2021-11

CONDITIONS: Strength Training
Keywords: eccentric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eccentric Training (Experimental): This Group will train on the KREHA for 20 Trainings
  Interventions: Other: eccentric arm-cranking training

INTERVENTIONS:
Other: eccentric arm-cranking training — Over the twenty training sessions, able-bodied participants will exercise on the KREHA device. An arm-crank has to be decelerated, which will be rotated by a prematurely defined revolution rate and training duration. During this intervention a certain power has to be applied. During the whole time of training a continous progression in power and training duration is applied

SUMMARY:
The new training device, the eccentric arm-crank, will be examined for its training effect by this project. That the training device can be used in athletes and patients with paraplegia in the future, the so-called "testing of the applicability of this concept" will be carried out during this study. Fourteen volunteer, healthy and trained people are first tested for their upper body performance, followed by a training phase over 20 trainings and at the and the performance data is collected again. The training intensity and duration is continuously increased during the training phase.

DETAILED DESCRIPTION:
At the beginning, the study design includes an familiarisation appointment with performance tests and training on the eccentric arm-crank device (KREHA). At least one week later, the first test sequence including a maximum strength test (bench press), magnetic resonance imaging (MRI) to determine the muscle cross-section area of the upper arm and a test to determine the anaerobic performance (Wingate test) is conducted. The second test sequence takes place one to three days later. This includes a handgrip strength test, an aerobic endurance test (ramp test on the arm crank ergometer with ergospirometry) and a further familiarisation training on the KREHA. The training phase starts within two weeks after the pre-tests have been completed. There are two to a maximum of three trainings per week. These take 30 to 60 minutes and take place on the KREHA device under the supervision of the study staff. The training phase lasts a maximum of twelve weeks (20 training sessions). The first test sequence is repeated five to eight days after the last workout. The second test sequence takes place at the same time interval as in the pre-tests.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age between 18 and 50 years
* experience in strength training
* trained (minimum two times a week)
* healthy
* adequately informed and confirmed per signature

Exclusion Criteria:

* findings during anamnesis of study doctor
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Upper body Performance | through study completion, an average of 20 weeks
  Peak Power - maximal reached power, generated during the 30sec Wingate arm-crank test

SECONDARY OUTCOMES:
Endurance Oxygen consumption | through study completion, an average of 20 weeks
  VO2peak [ml/min/kg] - Basic Endurance test (Ergospirometry, arm-crank)
Endurance Power | through study completion, an average of 20 weeks
  Wmax [W] - Basic Endurance test (Ergospirometry, arm-crank)
Upper body Mean Power | through study completion, an average of 20 weeks
  Mean Power [W] - Wingate Test (arm-crank)
Upper body Power - Time to Peak | through study completion, an average of 20 weeks
  Time to Peak [s] - Wingate Test (arm-crank)
Upper body Fatigue resistance | through study completion, an average of 20 weeks
  Fatigue Index [%]- Wingate Test (arm-crank)
Upper body Fatigue resistance | through study completion, an average of 20 weeks
  Fatigue Slope [W/s] - Wingate Test (arm-crank)
1RM bench press | through study completion, an average of 20 weeks
  One Repetition Maximum (1RM) [kg]- bench press
Grip Strength | through study completion, an average of 20 weeks
  Maximal Force that can be generated by pressing hand towards a fist [N]
Cross sectional muscle area | through study completion, an average of 20 weeks
  Cross sectional area of the upper arm is measured with MRI
Upper Arm Circumference | through study completion, an average of 20 weeks
  Circumference of the upper arm is measured with measuring tape

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No